CLINICAL TRIAL: NCT01113840
Title: Exercise Conditioning in Elderly Patients With Heart Failure
Brief Title: Prospective Aerobic Reconditioning Intervention Study
Acronym: PARIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.A.R.I.S. I and II; R01AG012257 (NIH); R01AG018915 (NIH)
Record Dates: First submitted 2010-04-29; First posted 2010-04-30 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure
Keywords: elderly; heart failure; exercise; diastolic dysfunction
MeSH Terms: conditions — Heart Failure; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Control group continues with their daily activity as they were prior to randomization. Receive bi-weekly follow-up phone calls to assess health status and encourage adherence with protocol.
  Interventions: Behavioral: Control
- Exercise (Active Comparator): Exercise classes three times per week in a controlled, supervised environment.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Exercise classes three times per week in a controlled, supervised environment.
  Arms: Exercise
Behavioral: Control — Control group continues daily life as prior to randomization.
  Arms: Control

SUMMARY:
The purpose of this study is :

* To determine if aerobic exercise conditioning can improve symptoms, cardiovascular function and quality of life in elderly patients with congestive heart failure.
* To describe the baseline clinical characteristics, cardiovascular function and neurohumoral function in elderly patients with congestive heart failure.
* To determine the specific cardiovascular and noncardiovascular mechanisms by which symptoms and quality of life may improve following exercise conditioning in elderly patients with congestive heart failure.

DETAILED DESCRIPTION:
In patients over age 65, cardiovascular disease accounts for the largest percentage of deaths, hospital days, doctor visits, and overall health care expenditures. In addition, heart failure is the most common discharge diagnosis in the elderly. Heart failure can be defined as a state in which cardiac output is insufficient to meet metabolic demands. This is most frequently manifested by symptoms of fatigue and dyspnea. Inherent in this definition is that symptoms may be increased or only occur during times when metabolic demand is increased, such as during exercise. As such, exercise intolerance is a hallmark of the heart failure syndrome. Exercise intolerance correlates not only with disease severity and also with subsequent mortality. Exercise tolerance can be objectively quantified during maximal symptom limited standardized exercise protocols by analysis of exercise time, workload, METS (metabolic equivalents), and oxygen consumption (V02)' These measures have appropriately become accepted as standards for functional assessment in this disorder as well as outcome measures following therapeutic interventions in HF. P.A.R.I.S. is a randomized, attention-controlled, single-blind trial of supervised aerobic exercise training in older patients with heart failure. The primary outcome is exercise capacity and the main secondary outcome is quality of life. Mechanistic outcomes were also examined. In PARIS, which focused on cardiac mechanisms, there were HFPEF and HFREF patients studied in parallel. In PARIS-II, there were only HFPEF patients which focused on vascular mechanisms.

Main outcomes have been reported (see citations below).

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 60 years of age
* Symptoms of congestive heart failure
* Able to understand and give informed consent

Exclusion Criteria:

* Age <60 years
* Does not have CHF
* Significant change in cardiac medication <3 weeks
* Myocardial infarction <3 weeks
* CABG surgery <3 months
* Angina pectoris not controlled during daily activity by pharmacological therapy or at <4 METS activity
* Sustained hypertension with systolic> 190 and diastolic> 110 on medications
* Valvular heart disease as the primary etiology of CHF
* Significant aortic stenosis
* Stroke of <3 months or with any physical restriction impairment that would prevent participation in exercise programs
* Chronic obstructive pulmonary disease on therapy that limits exercise duration
* Uncontrolled diabetes mellitus
* Active treatment for cancer or other noncardiovascular conditions with life expectancy less than three years
* Anemia "10 gms Hb)
* Renal insufficiency (cr >2.5 mg/dl)
* Psychiatric disease - uncontrolled major psychoses, depressions, dementia, or personality disorder
* Dementia - MMSE ~24 "22 for ~8th grade education)
* Lack of an acoustic window sufficient to allow definition of endocardial borders on the screening echocardiogram.
* Plans to leave area or be admitted to a nursing home within 2 years.
* Inability to walk at least 420 feet in 6 minutes without a cane or other assistive device.
* Inability to exercise at or near home.
* At the discretion of the clinical staff, it is believed that the participant cannot or will not complete the protocol because of frailty, illness, or other reason.
* Participation in a regular exercise regimen more than one time per week for at least twenty minutes per session; including but not limited to walking, swimming, weight lifting, golfing, or taking an exercise class.
* Inability to ambulate without cane or other assistive device during biomechanics testing or treadmill.
* Inability to attend at least fourteen weeks of the facility-based intervention

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 1993-07; Primary Completion 2004-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Peak exercise capacity | 16 weeks

SECONDARY OUTCOMES:
Quality of life | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dalane W Kitzman, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

REFERENCES:
- [Result] Kitzman DW, Little WC, Brubaker PH, Anderson RT, Hundley WG, Marburger CT, Brosnihan B, Morgan TM, Stewart KP. Pathophysiological characterization of isolated diastolic heart failure in comparison to systolic heart failure. JAMA. 2002 Nov 6;288(17):2144-50. doi: 10.1001/jama.288.17.2144. PMID 12413374
- [Result] Kitzman DW, Brubaker PH, Morgan TM, Stewart KP, Little WC. Exercise training in older patients with heart failure and preserved ejection fraction: a randomized, controlled, single-blind trial. Circ Heart Fail. 2010 Nov;3(6):659-67. doi: 10.1161/CIRCHEARTFAILURE.110.958785. Epub 2010 Sep 17. PMID 20852060
- [Result] Brubaker PH, Moore JB, Stewart KP, Wesley DJ, Kitzman DW. Endurance exercise training in older patients with heart failure: results from a randomized, controlled, single-blind trial. J Am Geriatr Soc. 2009 Nov;57(11):1982-9. doi: 10.1111/j.1532-5415.2009.02499.x. PMID 20121952
- [Result] John JM, Haykowsky M, Brubaker P, Stewart K, Kitzman DW. Decreased left ventricular distensibility in response to postural change in older patients with heart failure and preserved ejection fraction. Am J Physiol Heart Circ Physiol. 2010 Sep;299(3):H883-9. doi: 10.1152/ajpheart.00332.2010. Epub 2010 Jun 18. PMID 20562334
- [Result] Haykowsky MJ, Brubaker PH, John JM, Stewart KP, Morgan TM, Kitzman DW. Determinants of exercise intolerance in elderly heart failure patients with preserved ejection fraction. J Am Coll Cardiol. 2011 Jul 12;58(3):265-74. doi: 10.1016/j.jacc.2011.02.055. PMID 21737017
- [Result] Haykowsky MJ, Brubaker PH, Stewart KP, Morgan TM, Eggebeen J, Kitzman DW. Effect of endurance training on the determinants of peak exercise oxygen consumption in elderly patients with stable compensated heart failure and preserved ejection fraction. J Am Coll Cardiol. 2012 Jul 10;60(2):120-8. doi: 10.1016/j.jacc.2012.02.055. PMID 22766338
- [Result] Moore B, Brubaker PH, Stewart KP, Kitzman DW. VE/VCO2 slope in older heart failure patients with normal versus reduced ejection fraction compared with age-matched healthy controls. J Card Fail. 2007 May;13(4):259-62. doi: 10.1016/j.cardfail.2006.12.005. PMID 17517344
- [Result] Maldonado-Martin S, Brubaker PH, Kaminsky LA, Moore JB, Stewart KP, Kitzman DW. The relationship of a 6-min walk to VO(2 peak) and VT in older heart failure patients. Med Sci Sports Exerc. 2006 Jun;38(6):1047-53. doi: 10.1249/01.mss.0000222830.41735.14. PMID 16775543
- [Result] Brubaker PH, Joo KC, Stewart KP, Fray B, Moore B, Kitzman DW. Chronotropic incompetence and its contribution to exercise intolerance in older heart failure patients. J Cardiopulm Rehabil. 2006 Mar-Apr;26(2):86-9. doi: 10.1097/00008483-200603000-00007. No abstract available. PMID 16569976
- [Result] Brubaker PH, Marburger CT, Morgan TM, Fray B, Kitzman DW. Exercise responses of elderly patients with diastolic versus systolic heart failure. Med Sci Sports Exerc. 2003 Sep;35(9):1477-85. doi: 10.1249/01.MSS.0000084416.71232.EA. PMID 12972865
- [Result] Marburger CT, Brubaker PH, Pollock WE, Morgan TM, Kitzman DW. Reproducibility of cardiopulmonary exercise testing in elderly patients with congestive heart failure. Am J Cardiol. 1998 Oct 1;82(7):905-9. doi: 10.1016/s0002-9149(98)00502-5. PMID 9781977
- [Result] Kitzman DW, Brubaker PH, Herrington DM, Morgan TM, Stewart KP, Hundley WG, Abdelhamed A, Haykowsky MJ. Effect of endurance exercise training on endothelial function and arterial stiffness in older patients with heart failure and preserved ejection fraction: a randomized, controlled, single-blind trial. J Am Coll Cardiol. 2013 Aug 13;62(7):584-92. doi: 10.1016/j.jacc.2013.04.033. Epub 2013 May 9. PMID 23665370
- [Result] Haykowsky MJ, Herrington DM, Brubaker PH, Morgan TM, Hundley WG, Kitzman DW. Relationship of flow-mediated arterial dilation and exercise capacity in older patients with heart failure and preserved ejection fraction. J Gerontol A Biol Sci Med Sci. 2013 Feb;68(2):161-7. doi: 10.1093/gerona/gls099. Epub 2012 Apr 20. PMID 22522508
- [Result] Kitzman DW, Herrington DM, Brubaker PH, Moore JB, Eggebeen J, Haykowsky MJ. Carotid arterial stiffness and its relationship to exercise intolerance in older patients with heart failure and preserved ejection fraction. Hypertension. 2013 Jan;61(1):112-9. doi: 10.1161/HYPERTENSIONAHA.111.00163. Epub 2012 Nov 12. PMID 23150511
- [Result] Haykowsky MJ, Kouba EJ, Brubaker PH, Nicklas BJ, Eggebeen J, Kitzman DW. Skeletal muscle composition and its relation to exercise intolerance in older patients with heart failure and preserved ejection fraction. Am J Cardiol. 2014 Apr 1;113(7):1211-6. doi: 10.1016/j.amjcard.2013.12.031. Epub 2014 Jan 15. PMID 24507172